CLINICAL TRIAL: NCT01771822
Title: Cumulative Irritancy Patch Test (Cipt) of Ibuprofen 5% Topical Gel in Human Volunteers
Brief Title: Ibuprofen 5% Topical Gel CIPT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B3491004
Record Dates: First submitted 2012-12-05; First posted 2013-01-18 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Pain
Keywords: cumulative irritancy patch test (CIPT)
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Gels; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ibuprofen 5% topical gel (Experimental)
  Interventions: Drug: Ibuprofen 5% topical gel
- Topical gel vehicle (Experimental)
  Interventions: Drug: Topical gel vehicle
- Sodium lauryl sulfate 0.2% (Active Comparator)
  Interventions: Drug: Sodium lauryl sulfate 0.2%
- Sodium chloride solution 0.9% (saline) (Sham Comparator)
  Interventions: Drug: Sodium chloride solution 0.9% (saline)

INTERVENTIONS:
Drug: Ibuprofen 5% topical gel — 0.2 ml applied daily for 21 days over 3 weeks under occlusive conditions
  Arms: Ibuprofen 5% topical gel
Drug: Topical gel vehicle — 0.2 ml applied daily for 21 days over 3 weeks under occlusive conditions
  Arms: Topical gel vehicle
Drug: Sodium lauryl sulfate 0.2% — 0.2 ml applied daily for 21 days over 3 weeks under occlusive conditions
  Arms: Sodium lauryl sulfate 0.2%
Drug: Sodium chloride solution 0.9% (saline) — 0.2 ml applied daily for 21 days over 3 weeks under occlusive conditions
  Arms: Sodium chloride solution 0.9% (saline)

SUMMARY:
This study will determine the potential of Ibuprofen 5% Topical Gel and its vehicle gel to cause irritation after repeated topical application to the healthy skin of human subjects under controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and/or female subjects (to be confirmed by medical history) 18 years of age or older, female subjects of childbearing potential and males who are using an acceptable form of birth control, subjects who are free of any systemic or dermatologic disorder

Exclusion Criteria:

Have skin disease at the application site, not willing to stop use of systemic or topical analgesics, corticosteroids, or antihistamines, unwilling or unable to stop use of sunscreens, creams, or similar products on the back during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Assessment of local skin irritation at patch sites | Daily for 21 days, Days 2 through 22

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Days 1 through 22, + 28 days after last product administration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Carlstadt, New Jersey, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3491004&StudyName=Ibuprofen%205%25%20Topical%20Gel%20CIPT